CLINICAL TRIAL: NCT05614739
Title: FORAGER-1: A Phase 1, Open-Label, Multicenter Study of LOXO-435 (LY3866288) in Locally Advanced or Metastatic Solid Tumors Including Urothelial Cancer With FGFR3 Alterations
Brief Title: FORAGER-1: A Study of LOXO-435 (LY3866288) in Participants With Cancer With a Change in a Gene Called FGFR3
Acronym: FORAGER-1
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 18594; J4G-OX-JZVA (Other: Eli Lilly and Company); 2022-502755-59-00 (Other: EU CTR #); LOXO-FG3-22001 (Other: Eli Lilly and Company)
Record Dates: First submitted 2022-11-07; First posted 2022-11-14 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Urinary Bladder Neoplasms; Neoplasm Metastasis; Ureteral Neoplasms
Keywords: Bladder Cancer; Bladder Urothelial Carcinoma; Urinary Bladder Cancer; Urinary Tract Cancer; Renal Pelvis Cancer; Ureter Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms; Neoplasm Metastasis; Ureteral Neoplasms; Urologic Neoplasms | interventions — pembrolizumab; enfortumab vedotin

STUDY DESIGN:
Masking Description: Cohort A2 is randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Phase 1a: Cohort A1 LOXO-435 Monotherapy Dose Escalation (Experimental): LOXO-435 administered orally
  Interventions: Drug: LOXO-435
- Phase 1a: Cohort A2 LOXO-435 Monotherapy Dose Optimization (Experimental): LOXO-435 administered orally
  Interventions: Drug: LOXO-435
- Phase 1b: Cohort B1, B2, B4, and C1 LOXO-435 Monotherapy Dose Expansion (Experimental): LOXO-435 administered orally
  Interventions: Drug: LOXO-435
- Phase 1b: Cohort B3 LOXO-435 Plus Pembrolizumab (Experimental): LOXO-435 administered orally in combination with pembrolizumab administered intravenously (IV)
  Interventions: Drug: LOXO-435; Drug: Pembrolizumab
- Phase 1b: Cohort B5 LOXO-435 Plus Pembrolizumab Plus Enfortumab Vedotin (Experimental): LOXO-435 administered orally in combination with pembrolizumab administered IV and enfortumab vedotin administered IV
  Interventions: Drug: LOXO-435; Drug: Pembrolizumab; Drug: enfortumab vedotin

INTERVENTIONS:
Drug: LOXO-435 — Oral
  Other Names: LY3866288
Drug: Pembrolizumab — IV
  Arms: Phase 1b: Cohort B3 LOXO-435 Plus Pembrolizumab; Phase 1b: Cohort B5 LOXO-435 Plus Pembrolizumab Plus Enfortumab Vedotin
Drug: enfortumab vedotin — IV
  Arms: Phase 1b: Cohort B5 LOXO-435 Plus Pembrolizumab Plus Enfortumab Vedotin

SUMMARY:
The main purpose of this study is to learn more about the safety, side effects, and effectiveness of LOXO-435 by itself or when it is combined with other standard medicines that treat cancer. LOXO-435 may be used to treat cancer of the cells that line the urinary system and other solid tumor cancers that have a change in a particular gene (known as the FGFR3 gene). Participation could last up to 30 months (2.5 years) and possibly longer if the disease does not get worse.

DETAILED DESCRIPTION:
This is an open-label, multi-center, phase 1 study in participants with FGFR3-altered advanced solid tumor malignancy including metastatic urothelial cancer (UC). The study will be conducted in 2 phases: Phase 1a dose escalation (Cohort A1) and dose optimization (Cohort A2) and Phase 1b dose expansion. Phase 1a will assess safety, tolerability, and pharmacokinetics of LOXO-435 to determine the optimal dose for further expansion.

Phase 1b will include 6 dose expansion cohorts to evaluate the efficacy and safety of LOXO-435 as monotherapy or in combinations with pembrolizumab with or without enfortumab vedotin.

ELIGIBILITY:
Inclusion Criteria:

* Have solid tumor cancer with an FGFR3 pathway alteration on molecular testing in tumor or blood sample that is deemed as actionable

  * Cohort A1: Presence of an alteration in FGFR3 or its ligands
  * Cohort A2, B2, B3, and B5: Histological diagnosis of urothelial cancer (UC) that is locally advanced or metastatic with a qualifying FGFR3 genetic alteration
  * Cohorts B1 and B4: Histological diagnosis of urothelial cancer that is locally advanced or metastatic
  * Cohort C1: Must have histological diagnosis of a non-urothelial solid tumor malignancy that is locally advanced or metastatic with a qualifying FGFR3 genetic alteration
* Measurability of disease:

  * Cohort A1 and B3: Measurable or non-measurable disease as defined by Response Evaluation Criteria in Solid Tumors v 1.1 (RECIST v1.1)
  * Cohorts A2, B1, B2, B4, B5, and C1: Measurable disease required as defined by RECIST v1.1
* Have adequate tumor tissue sample available. Participants with inadequate tissue sample availability may still be considered for enrollment upon review
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 for Cohorts A1, A2, B3, and B5

  * Less than or equal to 2 for Cohorts B1, B2, B4, and C1
* Prior Systemic Therapy Criteria:

  * Cohort A1/C1: Participant has received all standard therapies for which the participant was deemed to be an appropriate candidate by the treating Investigator; OR the participant is refusing the remaining most appropriate standard of care treatment; OR there is no standard therapy available for the disease. There is no restriction on number of prior therapies.
  * Cohort A2, B2, B3 participants must have received at least one prior regimen, and cohorts B1 and B4 participants at least 2 prior regimens, in the locally advanced or metastatic setting
  * There is no restriction on number of prior therapies
* Cohort B5: Participants have not received prior systemic therapy for locally advanced or metastatic UC
* FGFR inhibitor specific requirements:

  * Cohort A1/A2/B3: Prior FGFR inhibitor treatment is permitted but not required
  * Cohort B1/B4: Participants must have been previously treated with erdafitinib
  * Cohort B2, B5, and C1: Participants must be FGFR inhibitor naïve

Exclusion Criteria:

* Participants with primary central nervous system (CNS) malignancy
* Untreated or uncontrolled CNS metastases
* Current evidence of corneal keratopathy or retinal disorder. Individuals with asymptomatic ophthalmic conditions may be eligible
* Any serious unresolved toxicities from prior therapy
* Significant cardiovascular disease
* Prolongation of the QT interval corrected for heart rate using Fridericia's formula (QTcF)
* Active uncontrolled systemic infection or other clinically significant medical conditions
* Participants who are pregnant, lactating, or plan to breastfeed during the study or within 6 months of the last dose of study treatment. Participants who have stopped breastfeeding may be enrolled

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 535 (Estimated)
Dates: Start 2023-01-12 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Phase 1a: To determine the recommended dose of LOXO-435: Safety, number of participants with dose-limiting toxicities (DLTs) | Minimum of the first 21-day cycle of LOXO-435 treatment
  Number of participants with DLTs
Phase 1b: To evaluate the preliminary antitumor activity of LOXO-435: Overall response rate (ORR) | Up to approximately 30 months or 2.5 years
  ORR per investigator assessed RECIST v1.1
Number of Participants with One or More Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Up to approximately 30 months or 2.5 years
  A summary of TEAEs and SAEs regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
To assess the pharmacokinetics (PK) of LOXO-435: Area under the concentration versus time curve (AUC) | Up to 2 months
  PK of LOXO-435: AUC
To assess the PK of LOXO-435: Minimum plasma concentration (Cmin) | Up to 2 months
  PK of LOXO-435: Cmin
To evaluate the preliminary antitumor activity of LOXO-435: Objective response rate (ORR) | Up to approximately 30 months or 2.5 years]
  ORR per investigator assessed RECIST 1.1
To evaluate the preliminary antitumor activity of LOXO-435: Duration of response (DoR) | Up to approximately 30 months or 2.5 years
  DOR per investigator assessed RECIST 1.1
To evaluate the preliminary antitumor activity of LOXO-435: Time to response (TTR) | Up to approximately 30 months or 2.5 years
  TTR
To evaluate the preliminary antitumor activity of LOXO-435: Progression-free survival (PFS) | Up to approximately 30 months or 2.5 years
  PFS per investigator assessed RECIST 1.1
To evaluate the preliminary antitumor activity of LOXO-435: Disease control rate (DCR) | Up to approximately 30 months or 2.5 years
  DCR per investigator assessed RECIST 1.1
To evaluate the preliminary antitumor activity of LOXO-435: Overall survival (OS) | Up to approximately 30 months or 2.5 years
  OS
Change from baseline in bladder-related symptoms, measured by Functional Assessment of Cancer Therapy - Bladder (FACT-Bl) subscale (BlCS) | Cycle 1 Day 1, Cycle 2 Day 1, and Cycle 3 Day 1 (28 day cycles)
  The BlCS has 12 items with a total score range of 0 to 48, with higher scores representing better bladder-related symptoms. A ≥ 4-point score change from baseline will be considered as clinically meaningful improvement in bladder-related symptoms
Change from baseline in physical function, measured by FACT- Physical Well-being Scale (PWB) subscale | Up to approximately 30 months or 2.5 years
  The PWB subscale has 7 items with a total score range of 0-28, with higher scores representing better physical function. A ≥ 3-point score change from baseline for a participant will be considered as clinically meaningful improvement in physical function.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (84):
- United States (42):
  - University of Arizona - Cancer Center, Tucson, Arizona
  - City of Hope, Duarte, California
  - University of California, Los Angeles (UCLA) - Division of Hematology-Oncology, Los Angeles, California
  - University of California - Irvine, Orange, California
  - University of California (UC) Davis Comprehensive Cancer Center, Sacramento, California
  - Stanford Cancer Center, Stanford, California
  - Advent Health, Orlando, Florida
  - Emory University Hospital, Atlanta, Georgia
  - The University of Chicago Medical Center (UCMC), Chicago, Illinois
  - Indiana University (IU) Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Johns Hopkins Kimmel Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Washington University in St. Louis, St Louis, Missouri
  - New York University (NYU), New York, New York
  - Weill Cornell Medicine, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Columbia University, New York, New York
  - David H. Koch Center for Cancer Care at Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester - Wilmot Cancer Institute, Rochester, New York
  - Montefiore Medical Center, The Bronx, New York
  - University of North Carolina (UNC) - Chapel Hill, Chapel Hill, North Carolina
  - University of Cincinnati Medical Center (UCMC), Cincinnati, Ohio
  - The Ohio State University (OSU), Columbus, Ohio
  - University of Oklahoma - Health Sciences Center, Oklahoma City, Oklahoma
  - Penn Medicine Lancaster General Hospital - Ann B. Barshinger Cancer Institute, Lancaster, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Sarah Cannon and HCA Research Institute, Nashville, Tennessee
  - Tennessee Oncology, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Southwestern, Dallas, Texas
  - Texas Oncology, P.A, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Vermont Medical Center, Burlington, Vermont
  - Inova Schar Cancer Institute, Falls Church, Virginia
- Australia (4):
  - St Vincent's Hospital, Darlinghurst
  - Calvary Mater Newcastle, Hunter Region, NSW
  - GenesisCare North Shore, St Leonards
  - Macquarie University, Sydney
- Canada (2):
  - Princess Margaret Hospital, Toronto
  - British Columbia Cancer Agency, Vancouver
- China (8):
  - Beijing Cancer hospital, Beijing
  - Beijing Hospital, Beijing
  - Sun Yat-Sen University- Cancer Center, Guangdong
  - Sir Run Run Shaw Hospital, School of Medicine, Zhejiang University, Hangzhou
  - Renji Hospital, Shanghai Jiaotong University School of Medicine, Shanghai
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin
  - First Affiliated Hospital of Medical College of Xian jiaotong University, Xi'an
  - Zhejiang Provincial People's Hospital, Zhejiang
- France (3):
  - Institut Bergonie, Bordeaux
  - Centre Leon Berard, Lyon
  - Institut Gustave Roussy, Villejuif
- Germany (3):
  - Universitaetsklinikum Schleswig-Holstein - Campus Luebeck, Lübeck
  - Klinikum der Technischen Universitaet Muenchen (TUM Klinikum), München
  - Universitaetsklinikum Tuebingen, Tübingen
- Israel (2):
  - Rabin Medical Center, Beilinson Hospital, Petah Tikva
  - Sheba Medical Center, Tel Litwinsky
- Italy (2):
  - IRCCS Ospedale San Raffaele, Milan
  - UOC Fase I - Fondazione Policlinico Universitario A. Gemelli IRCCS - Universita Cattolica del Sacro Cuore, Roma
- Japan (4):
  - National Cancer Center Hospital East, Chiba
  - Aichi Cancer Center Hospital, Nagoya
  - National Cancer Center Hospital, Tokyo
  - Cancer Institute Hospital of JFCR, Tokyo
- Erasmus MC, GE Rotterdam, Netherlands
- Norway (2):
  - Haukeland University Hospital, Bergen
  - Oslo University Hospital, Oslo
- South Korea (4):
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (5):
  - Institut Catala d'Oncologia - L'Hospitalet, Barcelona
  - Fundacion MD Anderson International Espana, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - South Texas Accelerated Research Therapeutics (START) Madrid - CIOCC, Madrid
  - Hospital Universitario Marques De Valdecilla, Santander
- United Kingdom (2):
  - The Christie NHS Foundation Trust, Manchester
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Study of LOXO-435 in Patients With Cancer With a Change in a Gene Called FGFR3 — https://trials.lilly.com/en-US/trial/367675